CLINICAL TRIAL: NCT00480025
Title: GSK1572932A Antigen-Specific Cancer Immunotherapeutic as Adjuvant Therapy in Patients With Resectable MAGE-A3 Positive Non-Small Cell Lung Cancer
Brief Title: GSK1572932A Antigen-Specific Cancer Immunotherapeutic as Adjuvant Therapy in Patients With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated following assessment of the lack of efficacy of the study product by the Independent Data monitoring Committee for the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109493; 2007-001283-73 (EudraCT Number); NCT00638105 (obsolete NCT alias)
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: ASCI; Immunotherapeutic; MAGRIT; Tumor antigen; Non-small-cell lung cancer; Adjuvant cancer therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK1572932 Group (Experimental): Patients received up to 13 doses of GSK1572932, 5 doses every 3 weeks followed by 8 doses every 12 weeks.
  Interventions: Biological: GSK1572932A Antigen-Specific Cancer Immunotherapeutic
- Placebo Group (Placebo Comparator): Patients received up to 13 doses of placebo, 5 doses every 3 weeks followed by 8 doses every 12 weeks.
  Interventions: Biological: Placebo Control

INTERVENTIONS:
Biological: GSK1572932A Antigen-Specific Cancer Immunotherapeutic — Intramuscular administration, 13 doses
  Arms: GSK1572932 Group
Biological: Placebo Control — Intramuscular administration, 13 doses
  Arms: Placebo Group

SUMMARY:
The purpose of this clinical trial is to demonstrate the benefit of the immunotherapeutic product GSK1572932A when given to patients with Non-Small Cell Lung Cancer, after removal of their tumor. A course of 13 injections will be administered over 27 months. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* Male or female patient with completely resected, pathologically proven stage IB, II or IIIA NSCLC.
* Written informed consent for MAGE-A3 expression screening on tumor biopsy has been obtained from the patient prior to shipment of the sample for expression testing (before or just after surgical resection), and written informed consent for the complete study has been obtained prior to the performance of any other protocol-specific procedure.
* Patient is ≥ 18 years of age at the time of signature of the first informed consent form.
* The patient's tumor shows expression of MAGE-A3 gene
* The surgical technique for resection of the patient's tumor is anatomical, involving at least a lobectomy or a sleeve lobectomy;
* The mediastinal lymph node sampling is done according to study protocol guidelines;
* The patient is free of metastasis, as confirmed by a negative baseline computer tomogram (CT scan) of the chest, upper abdomen and CT scan or MRI of the brain.

Other examinations should be performed as clinically indicated. Note that if randomization is taking place within 8 weeks after surgery, brain CT scans or brain MRI performed up to 4 weeks before surgery do not have to be repeated.

* ECOG performance status of 0, 1 or 2 at the time of randomization.
* Adequate bone-marrow reserve, adequate renal function and adequate hepatic function as assessed by standard laboratory criteria, and defined as:

Absolute neutrophil count ≥ 1.0 x 10E9/L Platelet count ≥ 75 x 10E9/L Serum creatinine ≤ 1.5 times the Upper Limit of Normal (ULN)

≤ 3.0 times the ULN if due to platinum adjuvant chemotherapy Total bilirubin ≤ 1.5 times the ULN Alanine transaminase (ALAT) ≤ 2.5 times the ULN

* If the patient is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post menopausal, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to administration of study treatment, have a negative pregnancy test and continue such precautions during all study treatment period and for 2 months after completion of the injection series.
* In the view of the investigator, the patient can and will comply with the requirements of the protocol.

Exclusion criteria

* The primary tumor was removed by segmentectomy or wedge resection.
* The patient shows any evidence of residual tumor after surgery.
* The patient has received any anti-cancer specific treatment, including radiotherapy, immunotherapy, chemotherapy or neo-adjuvant chemotherapy, except:

For the treatment of previous malignancies as allowed by the protocol (i.e., non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years), Administration of adjuvant platinum-based chemotherapy for the treatment of the current NSCLC is allowed between surgery and randomization.

* The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and highly likely to have been cured.
* History of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
* The patient has an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
* The patient requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents.

Note: The use of prednisone, or equivalent, <0.5 mg/kg/day (absolute maximum 40 mg/day), or inhaled corticosteroids for COPD or topical steroids is permitted.

* The patient has received a major organ allograft.
* The patient is known to be HIV-positive.
* The patient has an uncontrolled bleeding disorder.
* The patient has uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or uncontrolled arrhythmia at the time of enrolment.
* The patient needs home oxygenation.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures.
* The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has received any investigational or non-registered medicinal product other than the study medication within the 30 days preceding the first dose of study medication, or plans to receive such a drug during the study period.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2278 (Actual)
Dates: Start 2007-10-04 (Actual); Primary Completion 2013-12-06 (Actual); Study Completion 2014-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (499):
- United States (160):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Montebello, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Pleasant Hill, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, West Hollywood, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Torrington, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Alpharetta, Georgia
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Decatur, Illinois
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Harvey, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Munster, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Ashland, Kentucky
  - GSK Investigational Site, Hazard, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Lapeer, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Long Branch, New Jersey
  - GSK Investigational Site, Paramus, New Jersey
  - GSK Investigational Site, Armonk, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Danville, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Langhorne, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sayre, Pennsylvania
  - GSK Investigational Site, Wilkes-Barre, Pennsylvania
  - GSK Investigational Site, Willow Grove, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Cookeville, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Grapevine, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (9):
  - GSK Investigational Site, C.a.b.a., Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Cipolletti, Río Negro Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
- Australia (16):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Tweed Heads, New South Wales
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Chermside, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Richmond, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- Austria (6):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Wels
- Belgium (11):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Duffel
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Jette
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Namur
- Brazil (6):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Barretos, São Paulo
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (13):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Saint Catherines, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec
- China (14):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Harbin
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuhan
- Czechia (5):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Ústí nad Labem
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (4):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (35):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Beauvais
  - GSK Investigational Site, Béthune
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Elbeuf
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lorient
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Meaux
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Périgueux
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Grégoire
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Saint-Quentin
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Vannes
  - GSK Investigational Site, Villefranche-sur-Saône
- Germany (58):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Ebensfeld, Bavaria
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Frankfurt (Oder), Brandenburg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Braunschweig, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Oldenburg, Lower Saxony
  - GSK Investigational Site, Ostercappeln, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Lüdenscheid, North Rhine-Westphalia
  - GSK Investigational Site, Moers, North Rhine-Westphalia
  - GSK Investigational Site, Mülheim, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Troisdorf, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Waldbröl, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Zwickau, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Weißenfels, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Bad Berka, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bremen
  - GSK Investigational Site, Hamburg
- Greece (10):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chania
  - GSK Investigational Site, Heraklion
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Neo Faliro
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Piraeus
  - GSK Investigational Site, Pylaia
  - GSK Investigational Site, Thessaloniki
- Hong Kong (2):
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Shatin
- Hungary (11):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Deszk
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Mátraháza
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Pózva
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szombathely
- India (4):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
- Ireland (2):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
- Israel (6):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Zrifin
- Italy (25):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Lecco, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Orbassano (TO), Piedmont
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Monserrato, Sardinia
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Legnago, Veneto
  - GSK Investigational Site, Padua, Veneto
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Netherlands (5):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Nieuwegein
- Norway (2):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Trondheim
- Poland (14):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Chęciny
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Głuchołazy
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zakopane
- Russia (7):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Ufa
- GSK Investigational Site, Singapore, Singapore
- South Korea (3):
  - GSK Investigational Site, Kyunggi-do
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- Spain (13):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Leganés
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Sabadell
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Switzerland (6):
  - GSK Investigational Site, Aarau
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Bruderholz
  - GSK Investigational Site, Thun
  - GSK Investigational Site, Zurich
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Hat Yai
- Ukraine (9):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Vinnytsia
- United Kingdom (18):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Wythenshawe, Greater Manchester
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Bebington
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Inverness
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Maidstone
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4790

REFERENCES:
- [Background] Vansteenkiste JF, Cho BC, Vanakesa T, De Pas T, Zielinski M, Kim MS, Jassem J, Yoshimura M, Dahabreh J, Nakayama H, Havel L, Kondo H, Mitsudomi T, Zarogoulidis K, Gladkov OA, Udud K, Tada H, Hoffman H, Bugge A, Taylor P, Gonzalez EE, Liao ML, He J, Pujol JL, Louahed J, Debois M, Brichard V, Debruyne C, Therasse P, Altorki N. Efficacy of the MAGE-A3 cancer immunotherapeutic as adjuvant therapy in patients with resected MAGE-A3-positive non-small-cell lung cancer (MAGRIT): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2016 Jun;17(6):822-835. doi: 10.1016/S1470-2045(16)00099-1. Epub 2016 Apr 27. PMID 27132212
- [Background] Dizier B, Callegaro A, Debois M, Dreno B, Hersey P, Gogas HJ, Kirkwood JM, Vansteenkiste JF, Sequist LV, Atanackovic D, Goeman J, van Houwelingen H, Salceda S, Wang F, Therasse P, Debruyne C, Spiessens B, Brichard VG, Louahed J, Ulloa-Montoya F. A Th1/IFNgamma Gene Signature Is Prognostic in the Adjuvant Setting of Resectable High-Risk Melanoma but Not in Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 Apr 1;26(7):1725-1735. doi: 10.1158/1078-0432.CCR-18-3717. Epub 2019 Nov 15. PMID 31732522
- [Derived] Zhu J, Yuan Y, Wan X, Yin D, Li R, Chen W, Suo C, Song H. Immunotherapy (excluding checkpoint inhibitors) for stage I to III non-small cell lung cancer treated with surgery or radiotherapy with curative intent. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD011300. doi: 10.1002/14651858.CD011300.pub3. PMID 34870327
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109493 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2315 patients were screened towards participation in the study. For 3 of these subjects informed consent forms issues were reported, and thus only 2312 subjects were considered for analyses/results Out of these 2312 subjects, 2278 were enrolled in the study.
Pre-assignment Details: Out of the 2278 patients initially enrolled into the study, only 2272 patients received at least one dose of study treatment (1515 received GSK1572932 and 757 received placebo).
Period: Overall Study
Arm/Group | GSK1572932 Group | Placebo Group
Started | 1515 | 757
Completed | 763 | 388
Not Completed | 752 | 369
Not completed — Protocol Violation | 12 | 7
Not completed — Patients remaining ongoing at Data Lock | 101 | 55
Not completed — Disease Progression / Recurrence | 449 | 224
Not completed — Adverse Event | 44 | 12
Not completed — Other | 70 | 29
Not completed — SAE including intercurrent illness | 76 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1572932 Group | Placebo Group | Total
Number analyzed (Participants) | 1515 | 757 | 2272
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (8.96) | 63.4 (9.15) | 63.2 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370 | 179 | 549
  Male | 1145 | 578 | 1723
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 14 | 7 | 21
  Geographic ancestry: American Indian or Alaskan Native | 0 | 1 | 1
  Geographic ancestry: Asian - Central/South Asian heritage | 8 | 5 | 13
  Geographic ancestry: Asian - East Asian heritage | 195 | 112 | 307
  Geographic ancestry: Asian - Japanese heritage | 138 | 71 | 209
  Geographic ancestry: Asian - South East Asian heritage | 13 | 10 | 23
  Geographic ancestry: Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Geographic ancestry: White - Arabic//North African heritage | 7 | 9 | 16
  Geographic ancestry: White - Caucasian/European heritage | 1129 | 539 | 1668
  Geographic ancestry: Other | 11 | 1 | 12
  Geographic ancestry: Missing confirmed | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Person Year Rate (PYAR) as Regards Disease-free Survival (DFS) in the Overall Population
Description: DFS = time interval from randomization to 1st evidence of recurrence/death, if occurring before. All recurrence types were included, including local, regional & distant metastasis & 2nd primary lung cancer (i.e. local recurrence, defined as a tumor within same lung or at bronchial stump; regional recurrence, involving a clinically or radiologically manifest disease in mediastinum or supraclavicular nodes; & distant recurrence [any tumor arising in contralateral lung or outside hemithorax]). Deaths occurring without prior documentation of recurrence were considered as event & not censored. If no event occurred by time of analysis, time to event was censored at last assessment date of patient. New 1ry cancers outside lungs were not considered as event. PYAR= n (number of subjects reported with at least 1 event) divided by T (sum of follow-up period [in years] censored at 1st occurrence of event in group). Median DFS estimates were obtained non-parametrically by Kaplan-Meier method.
Time Frame: From administration of first dose of GSK1572932 study product/placebo solution to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as randomized included patients in the treatment group as allocated by the randomization system at the start of the study.
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
events/person-years | 0.17 | 0.168
Statistical Analysis 1: Comparison: GSK1572932 Group vs Placebo Group; Analysis compared DFS PYAR between groups for period from 1st treatment dose to DLP. A Cox model was used to evaluate treatment efficacy (TE). TE was calculated as PYAR in GSK1572932 Group (PYAR1) divided by PYAR in Placebo Group (PYAR2), and weighed for adjustment factors. This comparison in all patients (overall population) also included taking into account stratification by previous CT vs. No-CT treatment and weighing using randomization-minimization factors (RMF) as regressors; Test type: Superiority — RMF included: 1) Number of chemotherapy cycles received (1, 2 vs. 3, 4), if any; 2) Pathological stage of the disease (IB vs. II vs. IIIA); 3) Type of lymph-node sampling (minimal lymph-node sampling vs. systematic radical mediastinal lymphadenectomy); 4) ECOG performance status randomization (0, 1 vs. 2); 5) Smoking status ( 100 cigarettes a lifetime vs. > 100 cigarettes and current smoker vs. >100 cigarettes and past smoker); p = 0.7379, Regression, Cox — 2-sided p-value of Likelihood Ratio test from RMF-adjusted Cox regression, Efron method used to handle ties; Overall population objective reached if p-value < 2.56%/4% in absence/presence of statistically significant effect in the No-CT population; Treatment Efficacy = 1.024, 95% CI 2-sided [0.891 to 1.177]

2. Primary Outcome: Person Year Rate (PYAR) as Regards Disease-free Survival (DFS) in the No-CT Population
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Groups:
- GSK1572932 No-CT Group: Patients received up to 13 doses (D) of GSK1572932 ASCI, 5 Ds every 3 weeks followed by 8 Ds every 12 weeks. Patients in this sub-group consisted solely of patients who had not received adjuvant chemotherapy prior to randomization (No-CT Population).
- Placebo No-CT Group: Patients received up to 13 doses (D) of placebo, 5 Ds every 3 weeks followed by 8 Ds every 12 weeks. Patients in this sub-group consisted solely of patients who had not received adjuvant chemotherapy prior to randomization (No-CT Population).
Arm/Group | GSK1572932 No-CT Group | Placebo No-CT Group
Number analyzed (Participants) | 731 | 365
events/person-years | 0.169 | 0.178
Statistical Analysis 1: Comparison: GSK1572932 No-CT Group vs Placebo No-CT Group; Analysis compared DFS PYAR between groups for the period from 1st treatment dose to DLP. A Cox model was used to evaluate treatment efficacy (TE). TE was calculated as PYAR in GSK1572932 No-CT Group (PYAR1) divided by PYAR in Placebo No-CT Group (PYAR2) and weighed for adjustment factors. This comparison in all patients (overall population) also included taking into account weighing using randomization-minimization factors (RMF) as regressors; Test type: Superiority — RMF taken into account included: 1) Number of chemotherapy cycles received (1, 2 vs. 3, 4), if any; 2) Pathological stage of the disease (IB vs. II vs. IIIA); 3) Type of lymph-node sampling (minimal lymph-node sampling vs. systematic radical mediastinal lymphadenectomy); 4) ECOG performance status randomization (0, 1 vs. 2); 5) Smoking status ( 100 cigarettes a lifetime vs. > 100 cigarettes and current smoker vs. > 100 cigarettes and past smoker); p = 0.7572, Regression, Cox — 2-sided p-value of Likelihood Ratio test from RMF-adjusted Cox regression, Efron method used to handle ties; No-CT population objective reached if p-value < 2.56%/4% in absence/presence of statistically significant effect in the No-CT population; Treatment Efficacy = 0.97, 95% CI 2-sided [0.797 to 1.179]

3. Secondary Outcome: Person Year Rate (PYAR) as Regards Disease-free Survival (DFS) in the CT Population
Description: DFS = time interval from randomization to 1st evidence of recurrence/death, if occurring before. All recurrence types were included, including local, regional & distant metastasis & 2nd primary lung cancer (i.e. local recurrence, defined as a tumor within same lung or at bronchial stump; regional recurrence, involving a clinically or radiologically manifest disease in mediastinum or supraclavicular nodes; & distant recurrence [any tumor arising in contralateral lung or outside hemithorax]). Deaths occurring without prior documentation of recurrence were considered as event & not censored. If no event occurred by time of analysis, time to event was censored at last assessment date of patient. New 1ry cancers outside lungs were not considered as event. PYAR = n (number of subjects reported with at least 1 event) divided by T (sum of follow-up period [in years] censored at 1st occurrence of event in group). Median DFS estimates were obtained non-parametrically by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Groups:
- GSK1572932 CT Group: Patients received up to 13 doses (D) of GSK1572932, 5 Ds every 3 weeks followed by 8 Ds every 12 weeks. Patients in this sub-group consisted solely of patients who had received adjuvant chemotherapy prior to randomization (CT Population).
- Placebo CT Group: Patients received up to 13 doses (D) of placebo, 5 Ds every 3 weeks followed by 8 Ds every 12 weeks. Patients in this sub-group consisted solely of patients who had received adjuvant chemotherapy prior to randomization (CT Population).
Arm/Group | GSK1572932 CT Group | Placebo CT Group
Number analyzed (Participants) | 784 | 392
events/person-years | 0.172 | 0.158

4. Secondary Outcome: Person Year Rate (PYAR) as Regards Overall-survival (OS) in the Overall Population
Description: OS was defined as the time interval from randomization to the date of death, irrespective of the cause of death. Patients still alive were censored at the last visit they were known to be alive. PYAR = n (number of subjects reported with at least 1 event) divided by T (sum of follow-up period [in years] censored at 1st occurrence of event in group). Median OS estimates were obtained non-parametrically by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
events/person-years | 0.082 | 0.081

5. Secondary Outcome: Person Year Rate (PYAR) as Regards Overall-survival (OS) in the No-CT Population
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 No-CT Group | Placebo No-CT Group
Number analyzed (Participants) | 731 | 365
events/person-years | 0.084 | 0.086

6. Secondary Outcome: Person Year Rate (PYAR) as Regards Overall-survival (OS) in the CT Population
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 CT Group | Placebo CT Group
Number analyzed (Participants) | 784 | 392
events/person-years | 0.08 | 0.076

7. Secondary Outcome: Person Year Rate (PYAR) as Regards Lung-cancer Specific Survival (LCSS) in the Overall Population
Description: LCSS was defined as the time interval from randomization to the date of death due to lung cancer. Deaths due to other or unknown causes were censored at the date of death. PYAR = n (number of subjects reported with at least 1 event) divided by T (sum of follow-up period [in years] censored at 1st occurrence of event in group). Median OS estimates were obtained non-parametrically by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
events/person-years | 0.064 | 0.061

8. Secondary Outcome: Person Year Rate (PYAR) as Regards Lung-cancer Specific Survival (LCSS) in the No-CT Population
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 No-CT Group | Placebo No-CT Group
Number analyzed (Participants) | 731 | 365
events/person-years | 0.064 | 0.06

9. Secondary Outcome: Person Year Rate (PYAR) as Regards Lung-cancer Specific Survival (LCSS) in the CT Population
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 CT Group | Placebo CT Group
Number analyzed (Participants) | 784 | 392
events/person-years | 0.063 | 0.063

10. Secondary Outcome: Kaplan-Meier Estimate (KME) of 2, 3, 4 and 5-year as Regards Disease-free Survival (DFS) in the Overall Population
Description: DFS = time interval from randomization to 1st evidence of recurrence/death, if occurring before. All recurrence types were included, including local, regional & distant metastasis & 2nd primary lung cancer (i.e. local recurrence, defined as a tumor within same lung or at bronchial stump; regional recurrence, involving a clinically or radiologically manifest disease in mediastinum or supraclavicular nodes; & distant recurrence [any tumor arising in contralateral lung or outside hemithorax]). Deaths occurring without prior documentation of recurrence were considered as event & not censored. If no event occurred by time of analysis, time to event was censored at last assessment date of patient. New 1ry cancers outside lungs were not considered as event. Median DFS KMEs in % were obtained non-parametrically by Kaplan-Meier method and confidence intervals (CIs) calculated using the Greenwood formula for standard error computation.
Time Frame: KME assessed at 2, 3, 4 and 5-year (Y) post Dose 1 of treatment. Follow-up period was from administration of 1st dose of GSK1572932 study product/placebo solution to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent probability
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
percent probability
  DFS KME at 2Y - Overall Population | 65.57 [63.08 to 67.95] | 65.5 [61.94 to 68.81]
  DFS KME at 3Y - Overall Population | 59.97 [57.3 to 62.53] | 60.42 [56.62 to 64]
  DFS KME at 4Y - Overall Population | 56.72 [53.8 to 59.54] | 57.19 [53.07 to 61.1]
  DFS KME at 5Y - Overall Population | 51.73 [47.66 to 55.64] | 49.56 [42.87 to 55.88]

11. Secondary Outcome: Kaplan-Meier Estimate (KME) of 2, 3, 4 and 5-year as Regards Disease-free Survival (DFS) in the No-CT Population
Description: as for outcome 10
Time Frame: KME assessed at 2, 3, 4 and 5-year (Y) post Dose 1 of treatment Follow-up period was from administration of 1st dose of GSK1572932 study product/placebo solution to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent probability
Arm/Group | GSK1572932 No-CT Group | Placebo No-CT Group
Number analyzed (Participants) | 731 | 365
percent probability
  DFS KME at 2Y - No-CT Population | 66.03 [62.39 to 69.4] | 63.96 [58.72 to 68.72]
  DFS KME at 3Y - No-CT Population | 59.6 [55.7 to 63.27] | 57.62 [52.02 to 62.81]
  DFS KME at 4Y - No-CT Population | 55.4 [51.06 to 59.52] | 54.85 [48.98 to 60.33]
  DFS KME at 5Y - No-CT Population | 49.72 [43.44 to 55.67] | 44.59 [34.64 to 54.05]

12. Secondary Outcome: Kaplan-Meier Estimate (KME) of 2, 3, 4 and 5-year as Regards Disease-free Survival (DFS) in the CT Population
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent probability
Arm/Group | GSK1572932 CT Group | Placebo CT Group
Number analyzed (Participants) | 784 | 392
percent probability
  DFS KME at 2Y - CT Population | 65.17 [61.67 to 68.43] | 66.94 [61.98 to 71.41]
  DFS KME at 3Y - CT Population | 60.39 [56.68 to 63.89] | 63.09 [57.84 to 67.87]
  DFS KME at 4Y - CT Population | 58.17 [54.22 to 61.9] | 59.3 [53.33 to 64.76]
  DFS KME at 5Y - CT Population | 53.64 [48.28 to 58.7] | 54.8 [46.44 to 62.39]

13. Secondary Outcome: Person Year Rate (PYAR) as Regards Disease-free Specific Survival (DFSS) in the Overall Population
Description: DFSS was defined as the interval from randomization to the date of disease recurrence or death due to lung cancer. Patients who had died due to another cause than lung cancer were censored on their date of death and patients alive at the time of analysis were censored on the date of last assessment. Patients with no assessment post-randomization were censored on the date of randomization. PYAR = n (number of subjects reported with at least 1 event) divided by T (sum of follow-up period [in years] censored at 1st occurrence of event in group). Median DFS estimates were obtained non-parametrically by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
events/person-years | 0.159 | 0.154

14. Secondary Outcome: Person Year Rate (PYAR) as Regards Disease-free Specific Survival (DFSS) in the No-CT Population
Description: as for outcome 13
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 No-CT Group | Placebo No-CT Group
Number analyzed (Participants) | 731 | 365
events/person-years | 0.155 | 0.159

15. Secondary Outcome: Person Year Rate (PYAR) as Regards Disease-free Specific Survival (DFSS) in the CT Population
Description: as for outcome 13
Time Frame: Period of follow-up was from administration of first dose of GSK1572932 study product/placebo solution to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: as for outcome 1
Measure: Number; unit: events/person-years
Arm/Group | GSK1572932 CT Group | Placebo CT Group
Number analyzed (Participants) | 784 | 392
events/person-years | 0.162 | 0.149

16. Secondary Outcome: Number of Subjects Seropositive for Anti-Melanoma AntiGEn (MAGE)-A3 Antibodies (Anti-MAGE-A3 S+)
Description: A seropositive subject for anti-MAGE-A3 antibodies was a subject with anti-MAGE-A3 antibodies >= the seropositivity cut-off of 27 Enzyme-linked immunosorbent assay (ELISA) units per millilitre (EL.U/mL).
Time Frame: Pre-treatment (PRE), at Weeks (W) 6 and 12, at Months (M) 9, 12, 18 and 30 and at one year after treatment concluding time point, i.e. at follow-up visit 2 at W120 added of one year (At 12M post W120)
Population: The According-To-Protocol (ATP) population for immunogenicity including all evaluable patients (meeting all eligibility criteria, complying with protocol defined procedures and intervals, with no elimination criteria during the study) who received at least the 4 first doses and for whom data were available for the considered assay and time point.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1184 | 614
Participants
  Anti-MAGE-A3 S+, PRE | 105 | 53
  Anti-MAGE-A3 S+, W6: number analyzed (Participants) | 945 | 548
  Anti-MAGE-A3 S+, W6 | 929 | 43
  Anti-MAGE-A3 S+, W12: number analyzed (Participants) | 925 | 491
  Anti-MAGE-A3 S+, W12 | 921 | 42
  Anti-MAGE-A3 S+, M9: number analyzed (Participants) | 633 | 352
  Anti-MAGE-A3 S+, M9 | 631 | 30
  Anti-MAGE-A3 S+, M12: number analyzed (Participants) | 538 | 279
  Anti-MAGE-A3 S+, M12 | 536 | 19
  Anti-MAGE-A3 S+, M18: number analyzed (Participants) | 420 | 229
  Anti-MAGE-A3 S+, M18 | 419 | 15
  Anti-MAGE-A3 S+, M30: number analyzed (Participants) | 384 | 222
  Anti-MAGE-A3 S+, M30 | 383 | 17
  Anti-MAGE-A3 S+, at 12M post W120: number analyzed (Participants) | 76 | 47
  Anti-MAGE-A3 S+, at 12M post W120 | 75 | 5

17. Secondary Outcome: Number of Humoral Responders as Regards Anti-Melanoma AntiGEn (MAGE)-A3 Antibodies (Anti-MAGE-A3 HR)
Description: A seropositive/seronegative subject for anti-MAGE-A3 antibodies was a subject with anti-MAGE-A3 antibodies >=/< the seropositivity cut-off of 27 Enzyme-linked immunosorbent assay (ELISA) units per millilitre (EL.U/mL). A humoral responder as regards anti-MAGE-A3 antibodies was defined as 1) for initially seronegative patients, a patient with post-administration Anti-MAGE-A3 antibody concentration >= 27 EL.U/mL; 2) for initially seropositive patients: post-treatment administration antibody concentration >= 2 fold the pre-treatment antibody concentration.
Time Frame: At Weeks (W) 6 and 12, at Months (M) 9, 12, 18 and 30 and at one year after treatment concluding time point, i.e. at follow-up visit 2 at W120 added of one year (at 12M post W120)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 942 | 548
Participants
  Anti-MAGE-A3 HR, W6 | 922 | 10
  Anti-MAGE-A3 HR, W12: number analyzed (Participants) | 920 | 491
  Anti-MAGE-A3 HR, W12 | 916 | 15
  Anti-MAGE-A3 HR, M9: number analyzed (Participants) | 630 | 352
  Anti-MAGE-A3 HR, M9 | 627 | 13
  Anti-MAGE-A3 HR, M12: number analyzed (Participants) | 537 | 279
  Anti-MAGE-A3 HR, M12 | 534 | 6
  Anti-MAGE-A3 HR, M18: number analyzed (Participants) | 420 | 229
  Anti-MAGE-A3 HR, M18 | 417 | 7
  Anti-MAGE-A3 HR, M30: number analyzed (Participants) | 382 | 222
  Anti-MAGE-A3 HR, M30 | 380 | 8
  Anti-MAGE-A3 HR, at 12M post W120: number analyzed (Participants) | 76 | 47
  Anti-MAGE-A3 HR, at 12M post W120 | 75 | 3

18. Secondary Outcome: Number of Subjects Seropositive for Anti-protein D (PD) Antibodies (Anti-PD S+)
Description: A seropositive subject for anti-PD antibodies was a subject with anti-PD antibodies >= the seropositivity cut-off of 100 Enzyme-linked immunosorbent assay (ELISA) units per millilitre (EL.U/mL).
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1096 | 554
Participants
  Anti-PD S+, PRE | 381 | 210
  Anti-PD S+, W6: number analyzed (Participants) | 967 | 493
  Anti-PD S+, W6 | 958 | 195
  Anti-PD S+, W12: number analyzed (Participants) | 864 | 436
  Anti-PD S+, W12 | 860 | 176
  Anti-PD S+, M9: number analyzed (Participants) | 582 | 311
  Anti-PD S+, M9 | 580 | 133
  Anti-PD S+, M12: number analyzed (Participants) | 485 | 243
  Anti-PD S+, M12 | 483 | 101
  Anti-PD S+, M18: number analyzed (Participants) | 376 | 197
  Anti-PD S+, M18 | 375 | 77
  Anti-PD S+, M30: number analyzed (Participants) | 358 | 189
  Anti-PD S+, M30 | 357 | 75
  Anti-PD S+, at 12M post W120: number analyzed (Participants) | 78 | 46
  Anti-PD S+, at 12M post W120 | 77 | 17

19. Secondary Outcome: Number of Humoral Responders as Regards Anti-protein D (PD) Antibodies (Anti-PD HR)
Description: A seropositive/seronegative subject for anti-PD antibodies was a subject with anti-PD antibodies ≥/< the seropositivity cut-off of 100 Enzyme-linked immunosorbent assay (ELISA) units per millilitre (EL.U/mL). A humoral responder as regards anti-PD antibodies was defined as 1) for initially seronegative patients, a patient with post-administration anti-PD antibody concentration ≥ 100 EL.U/mL; 2) for initially seropositive patients: post-administration antibody concentration ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 962 | 490
Participants
  Anti-PD HR, W6 | 945 | 27
  Anti-PD HR, W12: number analyzed (Participants) | 859 | 432
  Anti-PD HR, W12 | 853 | 35
  Anti-PD HR, M9: number analyzed (Participants) | 579 | 307
  Anti-PD HR, M9 | 575 | 26
  Anti-PD HR, M12: number analyzed (Participants) | 482 | 240
  Anti-PD HR, M12 | 479 | 19
  Anti-PD HR, M18: number analyzed (Participants) | 374 | 194
  Anti-PD HR, M18 | 370 | 21
  Anti-PD HR, M30: number analyzed (Participants) | 354 | 186
  Anti-PD HR, M30 | 352 | 17
  Anti-PD HR, at 12M post W120: number analyzed (Participants) | 78 | 46
  Anti-PD HR, at 12M post W120 | 77 | 4

20. Secondary Outcome: Health-related Quality of Life (HQL) Scores
Description: HQL was assessed using the EQ-5D generic health state classification and valuation system. The number and percentage of patients with each score within each dimension of the EQ-5D questionnaire (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) were tabulated at each assessment for each group. Each of these scores can take 3 levels: no problem (level 1), moderate problem (level 2) or extreme problem (level 3). Resulting descriptive mean and standard deviation (SD) for the EQ-5D Utility Value (EQ-5D UV) were tabulated. Valid EQ-5D data were defined as questionnaires assessed 1) on day of and before treatment administration; or 2) on day after treatment administration for W0, W6, W12; or 3)during follow-up visits or at time of recurrence. The EQ-5D total score ranges from -0.016 (worst health state) to 1.000 (best health state).
Time Frame: At Week (W) 0 on day of treatment (DoT) (W0 DoT), W0 on day post treatment (DpT) (W0 DpT), W6 DoT, W6 DpT, W12 DoT, W12 DpT, Month (M) 6, M9, M12, M24, 6M post W120, at recurrence, and at 12M post W120
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 226 | 103
Scores on a scale
  EQ-5D UV, At W0 DoT | 0.83 (0.152) | 0.823 (0.189)
  EQ-5D UV, At W0 DpT: number analyzed (Participants) | 206 | 93
  EQ-5D UV, At W0 DpT | 0.788 (0.182) | 0.838 (0.177)
  EQ-5D UV, At W6 DoT: number analyzed (Participants) | 215 | 99
  EQ-5D UV, At W6 DoT | 0.837 (0.182) | 0.825 (0.191)
  EQ-5D UV, At W6 DpT: number analyzed (Participants) | 188 | 94
  EQ-5D UV, At W6 DpT | 0.798 (0.205) | 0.835 (0.176)
  EQ-5D UV, At W12 DoT: number analyzed (Participants) | 201 | 97
  EQ-5D UV, At W12 DoT | 0.848 (0.158) | 0.811 (0.236)
  EQ-5D UV, At W12 DpT: number analyzed (Participants) | 186 | 87
  EQ-5D UV, At W12 DpT | 0.841 (0.152) | 0.831 (0.211)
  EQ-5D UV, At M6: number analyzed (Participants) | 176 | 84
  EQ-5D UV, At M6 | 0.847 (0.182) | 0.825 (0.236)
  EQ-5D UV, At M9: number analyzed (Participants) | 173 | 81
  EQ-5D UV, At M9 | 0.84 (0.197) | 0.81 (0.219)
  EQ-5D UV, At M12: number analyzed (Participants) | 146 | 69
  EQ-5D UV, At M12 | 0.857 (0.166) | 0.824 (0.214)
  EQ-5D UV, At M24: number analyzed (Participants) | 102 | 50
  EQ-5D UV, At M24 | 0.855 (0.179) | 0.865 (0.145)
  EQ-5D UV, At 6M post W120: number analyzed (Participants) | 7 | 3
  EQ-5D UV, At 6M post W120 | 0.723 (0.298) | 0.679 (0.073)
  EQ-5D UV, At recurrence: number analyzed (Participants) | 41 | 14
  EQ-5D UV, At recurrence | 0.662 (0.343) | 0.785 (0.159)
  EQ-5D UV, At 12M post W120: number analyzed (Participants) | 16 | 5
  EQ-5D UV, At 12M post W120 | 0.753 (0.199) | 0.777 (0.395)

21. Secondary Outcome: Number of Patients With Abnormal Alanine Aminotransferase (ALT) Values by Maximum Grade
Description: The status of each patient as regards ALT laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1 and G2. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  ALT - SCR UNK; DLP G0 | 1 | 0
  ALT - SCR UNK; DLP G1 | 1 | 1
  ALT - SCR UNK; DLP G2 | 0 | 0
  ALT - SCR UNK; DLP G3 | 0 | 0
  ALT - SCR UNK; DLP G4 | 0 | 0
  ALT - SCR UNK; DLP UNK | 3 | 1
  ALT - SCR G0; DLP G0 | 1133 | 588
  ALT - SCR G0; DLP G1 | 162 | 77
  ALT - SCR G0; DLP G2 | 17 | 8
  ALT - SCR G0; DLP G3 | 7 | 7
  ALT - SCR G0; DLP G4 | 1 | 1
  ALT - SCR G0; DLP UNK | 113 | 37
  ALT - SCR G1; DLP G0 | 34 | 14
  ALT - SCR G1; DLP G1 | 32 | 17
  ALT - SCR G1; DLP G2 | 4 | 3
  ALT - SCR G1; DLP G3 | 1 | 2
  ALT - SCR G1; DLP G4 | 0 | 0
  ALT - SCR G1; DLP UNK | 4 | 1
  ALT - SCR G2; DLP G0 | 0 | 0
  ALT - SCR G2; DLP G1 | 1 | 0
  ALT - SCR G2; DLP G2 | 1 | 0
  ALT - SCR G2; DLP G3 | 0 | 0
  ALT - SCR G2; DLP G4 | 0 | 0
  ALT - SCR G2; DLP UNK | 0 | 0

22. Secondary Outcome: Number of Patients With Abnormal Alanine Aspartate Aminotransferase (AST) Values by Maximum Grade
Description: The status of each patient as regards AST laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1 and G2. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  AST - SCR UNK; DLP G0 | 12 | 4
  AST - SCR UNK; DLP G1 | 5 | 2
  AST - SCR UNK; DLP G2 | 0 | 0
  AST - SCR UNK; DLP G3 | 0 | 0
  AST - SCR UNK; DLP G4 | 0 | 0
  AST - SCR UNK; DLP UNK | 5 | 2
  AST - SCR G0; DLP G0 | 1170 | 579
  AST - SCR G0; DLP G1 | 136 | 84
  AST - SCR G0; DLP G2 | 6 | 4
  AST - SCR G0; DLP G3 | 8 | 5
  AST - SCR G0; DLP G4 | 2 | 1
  AST - SCR G0; DLP UNK | 111 | 37
  AST - SCR G1; DLP G0 | 26 | 19
  AST - SCR G1; DLP G1 | 25 | 16
  AST - SCR G1; DLP G2 | 5 | 2
  AST - SCR G1; DLP G3 | 0 | 1
  AST - SCR G1; DLP G4 | 0 | 0
  AST - SCR G1; DLP UNK | 2 | 1
  AST - SCR G2; DLP G0 | 0 | 0
  AST - SCR G2; DLP G1 | 0 | 0
  AST - SCR G2; DLP G2 | 0 | 0
  AST - SCR G2; DLP G3 | 1 | 0
  AST - SCR G2; DLP G4 | 0 | 0
  AST - SCR G2; DLP UNK | 1 | 0

23. Secondary Outcome: Number of Patients With Abnormal Alkaline Phosphatase (ALKP) Values by Maximum Grade
Description: The status of each patient as regards ALKP laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1 and G2. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  ALKP - SCR UNK; DLP G0 | 21 | 3
  ALKP - SCR UNK; DLP G1 | 0 | 0
  ALKP - SCR UNK; DLP G2 | 0 | 0
  ALKP - SCR UNK; DLP G3 | 1 | 0
  ALKP - SCR UNK; DLP G4 | 0 | 0
  ALKP - SCR UNK; DLP UNK | 5 | 3
  ALKP - SCR G0; DLP G0 | 1121 | 569
  ALKP - SCR G0; DLP G1 | 99 | 63
  ALKP - SCR G0; DLP G2 | 3 | 2
  ALKP - SCR G0; DLP G3 | 1 | 0
  ALKP - SCR G0; DLP G4 | 0 | 0
  ALKP - SCR G0; DLP UNK | 107 | 39
  ALKP - SCR G1; DLP G0 | 63 | 35
  ALKP - SCR G1; DLP G1 | 79 | 38
  ALKP - SCR G1; DLP G2 | 1 | 0
  ALKP - SCR G1; DLP G3 | 1 | 0
  ALKP - SCR G1; DLP G4 | 0 | 0
  ALKP - SCR G1; DLP UNK | 11 | 4
  ALKP - SCR G2; DLP G0 | 0 | 0
  ALKP - SCR G2; DLP G1 | 2 | 1
  ALKP - SCR G2; DLP G2 | 0 | 0
  ALKP - SCR G2; DLP G3 | 0 | 0
  ALKP - SCR G2; DLP G4 | 0 | 0
  ALKP - SCR G2; DLP UNK | 0 | 0

24. Secondary Outcome: Number of Patients With Abnormal Bilirubin (BIL) Values by Maximum Grade
Description: The status of each patient as regards BIL laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0) and G1. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  BIL - SCR UNK; DLP G0 | 9 | 2
  BIL - SCR UNK; DLP G1 | 1 | 0
  BIL - SCR UNK; DLP G2 | 0 | 0
  BIL - SCR UNK; DLP G3 | 0 | 0
  BIL - SCR UNK; DLP G4 | 0 | 0
  BIL - SCR UNK; DLP UNK | 4 | 2
  BIL - SCR G0; DLP G0 | 1275 | 661
  BIL - SCR G0; DLP G1 | 74 | 28
  BIL - SCR G0; DLP G2 | 11 | 9
  BIL - SCR G0; DLP G3 | 1 | 2
  BIL - SCR G0; DLP G4 | 1 | 0
  BIL - SCR G0; DLP UNK | 114 | 37
  BIL - SCR G1; DLP G0 | 10 | 5
  BIL - SCR G1; DLP G1 | 8 | 9
  BIL - SCR G1; DLP G2 | 5 | 1
  BIL - SCR G1; DLP G3 | 1 | 0
  BIL - SCR G1; DLP G4 | 0 | 0
  BIL - SCR G1; DLP UNK | 1 | 1

25. Secondary Outcome: Number of Patients With Abnormal Creatinine (CREA) Values by Maximum Grade
Description: The status of each patient as regards CREA laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1 and G2. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  CREA - SCR UNK; DLP G0 | 2 | 0
  CREA - SCR UNK; DLP G1 | 0 | 0
  CREA - SCR UNK; DLP G2 | 0 | 0
  CREA - SCR UNK; DLP G3 | 0 | 0
  CREA - SCR UNK; DLP G4 | 2 | 0
  CREA - SCR UNK; DLP UNK | 1139 | 577
  CREA - SCR G0; DLP G0 | 126 | 74
  CREA - SCR G0; DLP G1 | 9 | 3
  CREA - SCR G0; DLP G2 | 3 | 1
  CREA - SCR G0; DLP G3 | 1 | 0
  CREA - SCR G0; DLP G4 | 103 | 32
  CREA - SCR G0; DLP UNK | 27 | 14
  CREA - SCR G1; DLP G0 | 72 | 44
  CREA - SCR G1; DLP G1 | 11 | 6
  CREA - SCR G1; DLP G2 | 0 | 0
  CREA - SCR G1; DLP G3 | 1 | 0
  CREA - SCR G1; DLP G4 | 6 | 4
  CREA - SCR G1; DLP UNK | 0 | 0
  CREA - SCR G2; DLP G0 | 7 | 2
  CREA - SCR G2; DLP G1 | 6 | 0
  CREA - SCR G2; DLP G2 | 0 | 0
  CREA - SCR G2; DLP G3 | 0 | 0
  CREA - SCR G2; DLP G4 | 0 | 0
  CREA - SCR G2; DLP UNK | 0 | 0

26. Secondary Outcome: Number of Patients With Abnormal Haemoglobin (HGB) Values by Maximum Grade
Description: The status of each patient as regards HGB laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1, G2 and G3. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  HGB - SCR UNK; DLP G0 | 3 | 0
  HGB - SCR UNK; DLP G1 | 1 | 0
  HGB - SCR UNK; DLP G2 | 0 | 0
  HGB - SCR UNK; DLP G3 | 0 | 0
  HGB - SCR UNK; DLP G4 | 0 | 0
  HGB - SCR UNK; DLP UNK | 3 | 0
  HGB - SCR G0; DLP G0 | 534 | 274
  HGB - SCR G0; DLP G1 | 70 | 26
  HGB - SCR G0; DLP G2 | 9 | 5
  HGB - SCR G0; DLP G3 | 1 | 1
  HGB - SCR G0; DLP G4 | 0 | 2
  HGB - SCR G0; DLP UNK | 50 | 19
  HGB - SCR G1; DLP G0 | 342 | 187
  HGB - SCR G1; DLP G1 | 310 | 142
  HGB - SCR G1; DLP G2 | 17 | 14
  HGB - SCR G1; DLP G3 | 6 | 3
  HGB - SCR G1; DLP G4 | 2 | 0
  HGB - SCR G1; DLP UNK | 49 | 15
  HGB - SCR G2; DLP G0 | 29 | 30
  HGB - SCR G2; DLP G1 | 63 | 31
  HGB - SCR G2; DLP G2 | 12 | 3
  HGB - SCR G2; DLP G3 | 1 | 3
  HGB - SCR G2; DLP G4 | 1 | 0
  HGB - SCR G2; DLP UNK | 6 | 0
  HGB - SCR G3; DLP G0 | 2 | 0
  HGB - SCR G3; DLP G1 | 3 | 1
  HGB - SCR G3; DLP G2 | 1 | 1
  HGB - SCR G3; DLP G3 | 0 | 0
  HGB - SCR G3; DLP G4 | 0 | 0
  HGB - SCR G3; DLP UNK | 0 | 0

27. Secondary Outcome: Number of Patients With Abnormal Leukocytes (LEU) Values by Maximum Grade
Description: The status of each patient as regards LEU laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1, G2 and G3. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  LEU - SCR UNK; DLP G0 | 1 | 0
  LEU - SCR UNK; DLP G1 | 0 | 0
  LEU - SCR UNK; DLP G2 | 0 | 0
  LEU - SCR UNK; DLP G3 | 0 | 0
  LEU - SCR UNK; DLP G4 | 0 | 0
  LEU - SCR UNK; DLP UNK | 1 | 0
  LEU - SCR G0; DLP G0 | 1259 | 652
  LEU - SCR G0; DLP G1 | 45 | 29
  LEU - SCR G0; DLP G2 | 4 | 2
  LEU - SCR G0; DLP G3 | 2 | 0
  LEU - SCR G0; DLP G4 | 6 | 2
  LEU - SCR G0; DLP UNK | 98 | 32
  LEU - SCR G1; DLP G0 | 54 | 24
  LEU - SCR G1; DLP G1 | 21 | 5
  LEU - SCR G1; DLP G2 | 2 | 1
  LEU - SCR G1; DLP G3 | 0 | 0
  LEU - SCR G1; DLP G4 | 0 | 1
  LEU - SCR G1; DLP UNK | 4 | 0
  LEU - SCR G2; DLP G0 | 13 | 6
  LEU - SCR G2; DLP G1 | 3 | 2
  LEU - SCR G2; DLP G2 | 2 | 0
  LEU - SCR G2; DLP G3 | 0 | 0
  LEU - SCR G2; DLP G4 | 0 | 0
  LEU - SCR G2; DLP UNK | 0 | 0
  LEU - SCR G3; DLP G0 | 0 | 1
  LEU - SCR G3; DLP G1 | 0 | 0
  LEU - SCR G3; DLP G2 | 0 | 0
  LEU - SCR G3; DLP G3 | 0 | 0
  LEU - SCR G3; DLP G4 | 0 | 0
  LEU - SCR G3; DLP UNK | 0 | 0

28. Secondary Outcome: Number of Patients With Abnormal Lymphocytes (LYM) Values by Maximum Grade
Description: The status of each patient as regards LYM laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1, G2 and G3. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  LYM - SCR UNK; DLP G0 | 12 | 3
  LYM - SCR UNK; DLP G1 | 3 | 1
  LYM - SCR UNK; DLP G2 | 0 | 0
  LYM - SCR UNK; DLP G3 | 0 | 0
  LYM - SCR UNK; DLP G4 | 0 | 0
  LYM - SCR UNK; DLP UNK | 4 | 2
  LYM - SCR G0; DLP G0 | 999 | 518
  LYM - SCR G0; DLP G1 | 160 | 89
  LYM - SCR G0; DLP G2 | 40 | 16
  LYM - SCR G0; DLP G3 | 5 | 0
  LYM - SCR G0; DLP G4 | 0 | 0
  LYM - SCR G0; DLP UNK | 96 | 35
  LYM - SCR G1; DLP G0 | 47 | 27
  LYM - SCR G1; DLP G1 | 86 | 42
  LYM - SCR G1; DLP G2 | 15 | 4
  LYM - SCR G1; DLP G3 | 1 | 4
  LYM - SCR G1; DLP G4 | 2 | 0
  LYM - SCR G1; DLP UNK | 20 | 5
  LYM - SCR G2; DLP G0 | 3 | 1
  LYM - SCR G2; DLP G1 | 7 | 2
  LYM - SCR G2; DLP G2 | 4 | 3
  LYM - SCR G2; DLP G3 | 2 | 1
  LYM - SCR G2; DLP G4 | 0 | 0
  LYM - SCR G2; DLP UNK | 0 | 1
  LYM - SCR G3; DLP G0 | 4 | 1
  LYM - SCR G3; DLP G1 | 1 | 2
  LYM - SCR G3; DLP G2 | 3 | 0
  LYM - SCR G3; DLP G3 | 1 | 0
  LYM - SCR G3; DLP G4 | 0 | 0
  LYM - SCR G3; DLP UNK | 0 | 0

29. Secondary Outcome: Number of Patients With Abnormal Neutrophils (NEU) Values by Maximum Grade
Description: The status of each patient as regards NEU laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1, G2, G3 and G4. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  NEU - SCR UNK; DLP G0 | 12 | 3
  NEU - SCR UNK; DLP G1 | 0 | 0
  NEU - SCR UNK; DLP G2 | 0 | 0
  NEU - SCR UNK; DLP G3 | 0 | 0
  NEU - SCR UNK; DLP G4 | 0 | 0
  NEU - SCR UNK; DLP UNK | 1 | 2
  NEU - SCR G0; DLP G0 | 1200 | 625
  NEU - SCR G0; DLP G1 | 47 | 28
  NEU - SCR G0; DLP G2 | 1 | 3
  NEU - SCR G0; DLP G3 | 2 | 1
  NEU - SCR G0; DLP G4 | 3 | 1
  NEU - SCR G0; DLP UNK | 111 | 37
  NEU - SCR G1; DLP G0 | 56 | 23
  NEU - SCR G1; DLP G1 | 31 | 10
  NEU - SCR G1; DLP G2 | 3 | 1
  NEU - SCR G1; DLP G3 | 0 | 0
  NEU - SCR G1; DLP G4 | 0 | 0
  NEU - SCR G1; DLP UNK | 3 | 2
  NEU - SCR G2; DLP G0 | 32 | 16
  NEU - SCR G2; DLP G1 | 5 | 1
  NEU - SCR G2; DLP G2 | 2 | 2
  NEU - SCR G2; DLP G3 | 0 | 0
  NEU - SCR G2; DLP G4 | 0 | 0
  NEU - SCR G2; DLP UNK | 1 | 1
  NEU - SCR G3; DLP G0 | 3 | 1
  NEU - SCR G3; DLP G1 | 0 | 0
  NEU - SCR G3; DLP G2 | 0 | 0
  NEU - SCR G3; DLP G3 | 0 | 0
  NEU - SCR G3; DLP G4 | 0 | 0
  NEU - SCR G3; DLP UNK | 0 | 0
  NEU - SCR G4; DLP G0 | 1 | 0
  NEU - SCR G4; DLP G1 | 0 | 0
  NEU - SCR G4; DLP G2 | 1 | 0
  NEU - SCR G4; DLP G3 | 0 | 0
  NEU - SCR G4; DLP G4 | 0 | 0
  NEU - SCR G4; DLP UNK | 0 | 0

30. Secondary Outcome: Number of Patients With Abnormal Platelets (PLA) Values by Maximum Grade
Description: The status of each patient as regards PLA laboratory values at baseline (SCR) up to DLP was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were unknown (UNK), Grade 0 (G0), G1 and G3. CTC grade statuses reported at DLP were G0, G1, G2, G3, G4, and UNK.
Time Frame: From screening (SCR) to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  PLA - SCR UNK; DLP G0 | 1 | 1
  PLA - SCR UNK; DLP G1 | 0 | 0
  PLA - SCR UNK; DLP G2 | 0 | 0
  PLA - SCR UNK; DLP G3 | 0 | 0
  PLA - SCR UNK; DLP G4 | 0 | 0
  PLA - SCR UNK; DLP UNK | 1 | 0
  PLA - SCR G0; DLP G0 | 1275 | 648
  PLA - SCR G0; DLP G1 | 78 | 38
  PLA - SCR G0; DLP G2 | 6 | 2
  PLA - SCR G0; DLP G3 | 1 | 0
  PLA - SCR G0; DLP G4 | 7 | 2
  PLA - SCR G0; DLP UNK | 98 | 35
  PLA - SCR G1; DLP G0 | 22 | 16
  PLA - SCR G1; DLP G1 | 17 | 10
  PLA - SCR G1; DLP G2 | 2 | 4
  PLA - SCR G1; DLP G3 | 1 | 0
  PLA - SCR G1; DLP G4 | 0 | 0
  PLA - SCR G1; DLP UNK | 5 | 0
  PLA - SCR G3; DLP G0 | 1 | 1
  PLA - SCR G3; DLP G1 | 0 | 0
  PLA - SCR G3; DLP G2 | 0 | 0
  PLA - SCR G3; DLP G3 | 0 | 0
  PLA - SCR G3; DLP G4 | 0 | 0
  PLA - SCR G3; DLP UNK | 0 | 0

31. Secondary Outcome: Number of Patients With Any Adverse Events (AEs) and With AEs by Maximum Grade Reported - Up to Data Lock Point (DLP)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs reported are here below tabulated irrespective of grade, as well as graded by maximum grade reported according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. Maximum grade reported and tabulated were Grade 1 (G1), G2, G3, G4 and G5. Any here below is defined as irrespective of CTC grade reported.
Time Frame: Within the 31-day follow-up period post treatment administration, up to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants
  Patients with any AEs | 1369 | 556
  Patients with G1 AEs | 563 | 225
  Patients with G2 AEs | 560 | 209
  Patients with G3 AEs | 184 | 88
  Patients with G4 AEs | 49 | 26
  Patients with G5 AEs | 13 | 8

32. Secondary Outcome: Number of Patients With Serious Adverse Events (SAEs) - Up to Data Lock Point (DLP)
Description: A SAE is any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study subject, or was a Grade 4 AE according to CTC for Adverse Events, Version 3.0. Events part of natural course of lung cancer (i.e., disease progression, recurrence) were captured towards clinical efficacy assessment (CEA) and were not reported as SAEs. Death due to a progressive disease was similarly recorded towards CEA, but not as an SAE. However, if progression of lung cancer disease was greater than normally be expected, or if investigators considered that there was a causal relationship between treatment or protocol design/procedures and disease progression/ recurrence, then it was reported as SAE. Any new cancer (non-related to lung cancer) was reported as SAE.
Time Frame: From screening (SCR) up to data lock point (DLP) on 23 January 2014 (up to 5 years per patient)
Population: The Total Treated population - as treated included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1572932 Group | Placebo Group
Number analyzed (Participants) | 1515 | 757
Participants | 330 | 164

ADVERSE EVENTS:
Time Frame: From screening (Day 0) up to data lock point (DLP) on 23 January 2014, for up to 5 years per patient.
Arm/Group | GSK1572932 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 30/1515 | 17/757
Serious Adverse Events (participants affected / at risk) | 330/1515 | 164/757
Other Adverse Events (participants affected / at risk) | 1225/1515 | 300/757
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1572932 Group (N=1515) | Placebo Group (N=757)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 5 (5)
Peripheral artery thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 4 (4)
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder transitional cell carcinoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 3 (3) | 3 (3)
Death (General disorders) | 2 (2) | 3 (3)
Euthanasia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 2 (2)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Adams-stokes syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (6) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 3 (4)
Cardiac fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2)
Coronary artery disease (Cardiac disorders) | 3 (3) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (6) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (5)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 4 (7)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 2 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 7 (7) | 2 (2)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 2 (2)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (3) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Citrobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (2)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 2 (3)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 3 (3) | 1 (1)
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 2 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 4 (4) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 26 (27) | 15 (16)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 4 (4)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Q fever (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Rickettsiosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1572932 Group (N=1515) | Placebo Group (N=757)
Arthralgia (Musculoskeletal and connective tissue disorders) | 105 (161) | 31 (35)
Asthenia (General disorders) | 92 (199) | 26 (55)
Chills (General disorders) | 118 (249) | 7 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 131 (155) | 71 (80)
Decreased appetite (Metabolism and nutrition disorders) | 79 (112) | 28 (30)
Diarrhoea (Gastrointestinal disorders) | 76 (110) | 31 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 83 (91) | 47 (52)
Erythema (Skin and subcutaneous tissue disorders) | 120 (258) | 6 (6)
Fatigue (General disorders) | 243 (579) | 50 (85)
Headache (Nervous system disorders) | 129 (241) | 40 (50)
Influenza like illness (General disorders) | 198 (682) | 23 (39)
Injection site erythema (General disorders) | 104 (344) | 3 (3)
Injection site pain (General disorders) | 476 (1880) | 35 (73)
Injection site reaction (General disorders) | 273 (1368) | 14 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 183 (588) | 20 (23)
Nausea (Gastrointestinal disorders) | 108 (177) | 36 (45)
Pain (General disorders) | 237 (578) | 14 (26)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 125 (251) | 24 (29)
Pyrexia (General disorders) | 529 (1732) | 38 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.